CLINICAL TRIAL: NCT03080051
Title: Phase 0 Evaluation of [18F]MNI-952 as a Potential PET Radioligand for Imaging Tau Protein in the Brain of Patients With Progressive Supranuclear Palsy or Alzheimer's Disease Compared to Healthy Volunteers
Brief Title: Evaluation of [18F]MNI-952 as a Potential PET Radioligand for Imaging Tau Protein in the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-952
Record Dates: First submitted 2017-01-12; First posted 2017-03-15 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Progressive Supranuclear Palsy; Alzheimer Disease; Healthy Volunteers
Keywords: PSP; AD; HV
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Alzheimer Disease | interventions — florbetapir

ARMS (1):
- [18F]MNI-952 (Experimental): To evaluate [18F]MNI-952 (also known as [18F]UCB-K), a tau targeted PET radioligand.
  Interventions: Drug: [18F]MNI-952; Drug: [18F]Florbetapir

INTERVENTIONS:
Drug: [18F]MNI-952 — Subjects will undergo PET imaging using [18F]MNI-952, a PET radioligand for imaging tau.
  Other Names: [18F]UCB-K
Drug: [18F]Florbetapir — Subjects with Alzheimer's disease will receive a [18F]florbetapir scan to compare distribution of tau in the brain compared to that of [18F]MNI-952.

SUMMARY:
The overall goal of this imaging trial is to evaluate [18F]MNI-952 (also known as [18F]UCB-K), a tau targeted PET radioligand.

DETAILED DESCRIPTION:
The overall goal of this imaging trial is to evaluate [18F]MNI-952 (also known as [18F]UCB-K), a tau targeted PET radioligand.

* To characterize [18F]MNI-952, a PET radioligand for imaging tau.
* To visually and quantitatively assess brain uptake and pharmacokinetics of [18F]MNI-952, a PET imaging marker for tau pathology in individuals with Progressive Supranuclear Palsy (PSP) or Alzheimer's disease (AD) and compare with healthy volunteers (HV).
* To evaluate the safety of a single injection of [18F]MNI-952.
* To compare the distribution of tau (using [18F]MNI-952) and Aâ (using florbetapir) in AD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for study duration and for 90 days following participation.
* Willing and able to cooperate with study procedures

Inclusion Criteria for healthy volunteer subjects:

* Males and females aged <55 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MNI-952 imaging visit.
* No neurologic impairment as judged by the investigator
* No family history of Alzheimer's disease or neurological disease associated with dementia
* Have a CDR score=0

Inclusion Criteria for subjects with a diagnosis of probable Alzheimer's disease (AD):

* Males and females aged between 50 and 90 years.
* Have probable Alzheimer's disease, based on the NINCDS/ADRDA and DSM-IV criteria.
* Have a CDR score of 0.5 or greater at screening.
* Have an MMSE score ≤ 28.
* Have a screening [18F]florbetapir PET imaging demonstrating amyloid binding based on qualitative (visual read)
* A brain MRI that supports a diagnosis of AD, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 30 days before the screening visit
* The subject has an appropriate caregiver capable of accompanying subject, if necessary.
* Signed and dated written informed consent obtained from the subject and/or the subject's legally authorized representative or caregiver (if applicable).

Inclusion Criteria for subjects with a diagnosis of probable Progressive Supranuclear Palsy (PSP):

* Males and females aged 50 to 90 years.
* Has a clinical diagnosis of PSP based on the NINDS and Society for PSP criteria (Litvan, et al 1996).
* Have screening DaTSCAN SPECT imaging demonstrating evidence of dopamine transporter deficit based on qualitative (visual) read.
* A brain MRI that supports a diagnosis of PSP, with no evidence of focal disease or MRI exclusion criteria.
* Medications taken for symptomatic treatment of PSP must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* The subject has an appropriate caregiver capable of accompanying subject, if necessary.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).

Exclusion Criteria:

* Current or prior history of any alcohol or drug abuse.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Subject has received an investigational drug or device within 30 days of screening
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines.
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: Findings of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Exclusion criteria for subjects with AD:

* Has received treatment that targeted amyloid-β or tau within the last 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Tracer uptake will be evaluated in regions of interest for analysis of regional [18F]MNI-952 binding/uptake and expressed in SUV by using established methods for normalization for 2 PSP, 2 AD, and 2 HV subjects. | 1 year
  Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MNI-952.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Madonia, PA-C, Principal Investigator — Molecular NeuroImaging
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- See also: Related Info — https://mnimaging.com/